CLINICAL TRIAL: NCT05584813
Title: Randomized Controlled Trial for Evaluation of Colour Vision Impairment During Acute Hypobaric Hypoxia in Aviation Medicine
Brief Title: Colour Vision Impairment During Acute Hypobaric Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DRU-COLOR-KOELN
Record Dates: First submitted 2022-09-27; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Hypoxia, Altitude
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Five different Groups were analyzed:
  * ground control binocular (n=12, Bi/GC)
  * ground control monocular (n=11, Mo/GC)
  * 10,000 ft, 60 min, monocular (n=10, Mo/60/10,000)
  * 15,000 ft, 15 min, binocular (n=11, Bi/15/15,000)
  * 15,000 ft, 60 min, monocular (n=10, Mo/60/15,000)
Who Masked: Participant
Masking Description: Volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ground control binocular (No Intervention): Intervention: pressure chamber environment Procedures: Colour vision tests were performed under normoxia with both eyes three times in a row for appropriate comparability to the simulated flight stages pre-peri-post hypoxia in the intervention groups
- ground control monocular (No Intervention): Intervention: pressure chamber environment Procedures: Colour vision tests were performed under normoxia with one eye at a time three times in a row for appropriate comparability to the simulated flight stages pre-peri-post hypoxia in the intervention groups
- 10,000 ft, 60 min, monocular pre-peri-post (Experimental): Intervention: Hypoxia equivalent to an altitude of 10.000 ft. for 60 minutes
  Procedures: Colour vision tests were performed with one eye at a time, thereby:
  * pre intervention with no hypoxia administered
  * during intervention with hypoxia equivalent to an altitude of 10.000 ft. for 60 minutes
  * post intervention with no hypoxia administered
  Interventions: Other: Hypobaric Hypoxia
- 15,000 ft, 15 min, binocular (Experimental): Intervention: Hypoxia equivalent to an altitude of 15.000 ft. for 15 minutes
  Procedures: Colour vision tests were performed with both eyes, thereby:
  * pre intervention with no hypoxia administered
  * during intervention with hypoxia equivalent to an altitude of 15000 ft. for 15 minutes
  * post intervention with no hypoxia administered
  Interventions: Other: Hypobaric Hypoxia
- 15,000 ft, 60 min, monocular (Experimental): Intervention: Hypoxia equivalent to an altitude of 15.000 ft. for 60 minutes
  Procedures: Colour vision tests were performed with one eye at a time, thereby:
  * pre intervention with no hypoxia administered
  * during intervention with hypoxia equivalent to an altitude of 15.000 ft. for 60 minutes
  * post intervention with no hypoxia administered
  Interventions: Other: Hypobaric Hypoxia

INTERVENTIONS:
Other: Hypobaric Hypoxia — The Waggoner Computerized Color Vision Test (WCCVT) and the Waggoner D-15 (WC-D15) were performed by 54 healthy volunteers in a decompression chamber.
  Arms: 10,000 ft, 60 min, monocular pre-peri-post; 15,000 ft, 15 min, binocular; 15,000 ft, 60 min, monocular

SUMMARY:
This study analyses the impairment of colour vision during hypobaric hypoxia in volunteers of different groups.

DETAILED DESCRIPTION:
This study analyses the impairment of colour vision during hypobaric hypoxia in volunteers of different groups.

Five different Groups were analysed:

* ground control binocular (n=12, Bi/GC)
* ground control monocular (n=11, Mo/GC)
* 10,000 ft, 60 min, monocular (n=10, Mo/60/10,000)
* 15,000 ft, 15 min, binocular (n=11, Bi/15/15,000)
* 15,000 ft, 60 min, monocular (n=10, Mo/60/15,000)

ELIGIBILITY:
Inclusion Criteria:

* volunteers from 18 years old

Exclusion Criteria:

* cardiovascular, pulmonary, neurological, or ear, nose, and throat disease
* pregnant or suffering from cold symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Colour vision pre hypoxia monocular/binocular Waggoner CCVT | Assessment was conducted 15 minutes before the start of the hypoxia intervention and the number of correctly identified plates in the Waggoner CCVT was collected
  Waggoner CCVT was administered in the pressure chamber pre hypoxia intervention, thereby the following parameters were collected:
  - the number of correctly identified plates in the Waggoner CCVT
  as of the study arm "15,000 ft, 15 min, binocular" the colour vision tests were performed binocularly
  as of the study arms "15,000 ft, 60 min, monocular" and "10,000 ft, 60 min, monocular" the colour vision tests were performed monocularly
  Time Frame - additional info:
  - depending on the time the subjects took for the colour vision tests, the time between the end of the pre-test and the onset of hypoxia was slightly variable
Colour vision pre hypoxia monocular/binocular D15 | Assessment was conducted 15 minutes before the start of the hypoxia intervention and S-Index, C-Index and TES in the Waggoner D15 were collected
  Waggoner D15 was administered in the pressure chamber pre hypoxia intervention, thereby the following parameters were collected:
  - S-Index, C-Index and TES in the Waggoner D15
  as of the study arm "15,000 ft, 15 min, binocular" the colour vision tests were performed binocularly
  as of the study arms "15,000 ft, 60 min, monocular" and "10,000 ft, 60 min, monocular" the colour vision tests were performed monocularly
  Time Frame - additional info: depending on the time the subjects took for the colour vision tests, the time between the end of the pre-test and the onset of hypoxia was slightly variable
Colour vision during hypoxia monocular/binocular Waggoner CCVT | Assessment was conducted immediately or 45 minutes after induction of hypoxia and the number of correctly identified plates in the Waggoner CCVT was collected
  Waggoner CCVT was administered in the pressure chamber during hypoxia intervention, thereby the following parameters were collected:
  - the number of correctly identified plates in the Waggoner CCVT
  as of the study arm "15,000 ft, 15 min, binocular" the colour vision tests were performed binocularly
  as of the study arms "15,000 ft, 60 min, monocular" and "10,000 ft, 60 min, monocular" the colour vision tests were performed monocularly
  Time Frame - additional info:
  * as of the study arm "15,000 ft, 15 min, binocular" assessment was conducted immediately after onset of hypoxia
  * as of the study arms "15,000 ft, 60 min, monocular" and "10,000 ft, 60 min, monocular" assessment was conducted 45 minutes after onset of hypoxia
  * depending on the time the subjects took for the colour vision tests, the time between the end of the peri-test and the end of hypoxia was slightly variable
Colour vision during hypoxia monocular/binocular D15 | Assessment was conducted immediately or 45 minutes after induction of hypoxia and S-Index, C-Index and TES in the Waggoner D15 were collected
  Waggoner D15 was administered in the pressure chamber during hypoxia intervention, thereby the following parameters were collected:
  - S-Index, C-Index and TES in the Waggoner D15
  as of the study arm "15,000 ft, 15 min, binocular" the colour vision tests were performed binocularly
  as of the study arms "15,000 ft, 60 min, monocular" and "10,000 ft, 60 min, monocular" the colour vision tests were performed monocularly
  Time Frame - additional info:
  * as of the study arm "15,000 ft, 15 min, binocular" assessment was conducted immediately after onset of hypoxia
  * as of the study arms "15,000 ft, 60 min, monocular" and "10,000 ft, 60 min, monocular" assessment was conducted 45 minutes after onset of hypoxia
  * depending on the time the subjects took for the colour vision tests, the time between the end of the peri-test and the end of hypoxia was slightly variable
Colour vision after hypoxia monocular/binocular Waggoner CCVT | Assessment was conducted immediately after hypoxia and the number of correctly identified plates in the Waggoner CCVT was collected
  Waggoner CCVT was administered in the pressure chamber post hypoxia intervention, thereby the following parameters were collected:
  - the number of correctly identified plates in the Waggoner CCVT
  as of the study arm "15,000 ft, 15 min, binocular" the colour vision tests were performed binocularly
  as of the study arms "15,000 ft, 60 min, monocular" and "10,000 ft, 60 min, monocular" the colour vision tests were performed monocularly
  Time Frame - additional info:
  * as of the study arm "15,000 ft, 15 min, binocular" assessment was conducted immediately after 15min of hypoxia
  * as of the study arms "15,000 ft, 60 min, monocular" and "10,000 ft, 60 min, monocular" assessment was conducted immediately after 60 minutes of hypoxia
Colour vision after hypoxia monocular/binocular D15 | Assessment was conducted immediately after hypoxia and S-Index, C-Index and TES in the Waggoner D15 were collected
  Waggoner D15 was administered in the pressure chamber post hypoxia intervention, thereby the following parameters were collected:
  - S-Index, C-Index and TES in the Waggoner D15
  as of the study arm "15,000 ft, 15 min, binocular" the colour vision tests were performed binocularly
  as of the study arms "15,000 ft, 60 min, monocular" and "10,000 ft, 60 min, monocular" the colour vision tests were performed monocularly
  Time Frame - additional info:
  * as of the study arm "15,000 ft, 15 min, binocular" assessment was conducted immediately after 15min of hypoxia
  * as of the study arms "15,000 ft, 60 min, monocular" and "10,000 ft, 60 min, monocular" assessment was conducted immediately after 60 minutes of hypoxia
Colour vision without hypoxia monocular/binocular Waggoner CCVT | Assessment was coducted independently of hypoxia three times in a row with a 1 minute break in between each test and the number of correctly identified plates in the Waggoner CCVT was collected
  Waggoner CCVT was administered three times in a row without hypoxia, thereby the following parameters were collected:
  - the number of correctly identified plates in the Waggoner CCVT
  as of the study arm "ground control binocular" the colour vision tests were performed binocularly
  as of the study arm "ground control monocular" the colour vision tests were performed monocularly
  Time Frame - additional info:
  - depending on the time the subjects took for each of the colour vision tests, total duration of all 3 test sequences can differ slightly
Colour vision without hypoxia monocular/binocular D15 | Assessment was coducted independently of hypoxia three times in a row with a 1 minute break in between each test, and S-Index, C-Index and TES in the Waggoner D15 were collected
  Waggoner D15 was administered three times in a row without hypoxia, thereby the following parameters were collected:
  - S-Index, C-Index and TES in the Waggoner D15
  as of the study arm "ground control binocular" the colour vision tests were performed binocularly
  as of the study arm "ground control monocular" the colour vision tests were performed monocularly
  Time Frame - additional info:
  - depending on the time the subjects took for each of the colour vision tests, total duration of all 3 test sequences can differ slightly

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Hinkelbein, Prof., Study Chair — University Hospital Cologne
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany